CLINICAL TRIAL: NCT02653027
Title: A Study of the Effect of Combination Lumacaftor and Ivacaftor on Glucose Tolerance in Persons With Cystic Fibrosis Who Are Homozygous for the Phe508del Cystic Fibrosis Transmembrane Conductance Regulator Mutation.
Brief Title: Effect of Lumacaftor-ivacaftor on Glucose Handling and Tolerance in Cystic Fibrosis Phe508del
Acronym: LIGHT-CF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Potential subjects were already on the combination therapy.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jose C. Florez, MD, PhD, Chief of the Diabetes Unit, Associate Professor Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2015P001811
Record Dates: First submitted 2016-01-07; First posted 2016-01-12 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Cystic Fibrosis
Keywords: Genetics
MeSH Terms: conditions — Diabetes Mellitus; Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumacaftor Ivacaftor (Experimental): Subjects will get an OGTT before and after starting the combination therapy lumacaftor-ivacaftor.
  Interventions: Drug: Lumacaftor-ivacaftor; Other: OGTT

INTERVENTIONS:
Drug: Lumacaftor-ivacaftor — Subjects who are planning on starting the combination therapy (lumacaftor-ivacaftor) will participate in OGTTs before and after starting the medication.
  Other Names: Orkambi
Other: OGTT — A subject is given an oral glucose load and insulin and glucose measurements are taken at specified time periods.
  Other Names: Oral Glucose tolerance test

SUMMARY:
The purpose of this research study is to find out if the combined therapy lumacaftor-ivacaftor effects how people with cystic fibrosis respond to an oral glucose tolerance test, a test for diabetes.

DETAILED DESCRIPTION:
This is a single center, open label study with crossover in patients with Cystic Fibrosis (CF). Patients will have 2-3 visits at the Diabetes Center at Massachusetts General Hospital (MGH).

The participants will have been previously screened clinically to make sure they are candidates for starting the combination drug, lumacaftor-ivacaftor. These patients will be contacted prior to their first visit to discuss enrollment in the study.

At the first study visit (Visit 1), the participant will come to the Diabetes Center after an overnight fast of at least 8 hours. The following will occur at this study visit: informed consent; brief medical history; weight and height; vital signs and blood pressure; blood draw for DNA extraction, and an extra research tube for storage; administration of 75g Glucola load as per a standard oral glucose tolerance test (OGTT) protocol; and blood work for glucose and insulin at 30, 60, 90 and 120 minutes after the glucose load. This will be scheduled at a time that is convenient to the patient, with an attempt to coordinate with the patient's visit to the CF clinic prior to starting lumacaftor-ivacaftor combination drug.

At the 2nd study visit (Visit 2), which will take place 3 months after starting the combination drug, the participant will again come to the Diabetes Center after an overnight fast of at least 8 hours. The participant will undergo a second OGTT as in the first visit. The 3rd study visit (Visit 3) will be 6 months after initiation of the drug, and will have a repeat administration of an OGTT. If a participant starts the combination drug before enrolling in the study, he/she can still participate in the study as long as he or she has had a clinical OGTT performed within 6 months of starting the combination drug. In these cases, the informed consent, brief medical history, weight and height and vital signs and blood pressure, as well as blood draw for DNA will occur on the Visit 2, which will be the first study visit for these participants. If a clinical OGTT had been performed prior to but within 6 months of starting the combination therapy, this OGTT can be used in analysis of the data, although will not have the full amount of data as the study OGTT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or greater
2. Patients diagnosed with CF, genotype homozygous PheDel508
3. Subject is planning on starting lumacaftor-ivacaftor for clinical reasons, with no contraindication for starting the drug* OR subject is taking combination drug and had an OGTT done at a partners facility in the 6 months prior to initiating the drug.

   * Contraindications for taking drug include abnormal liver enzyme tests, renal dysfunction, pregnancy or nursing mothers

Exclusion Criteria:

1. Currently taking any medications for diabetes (including oral or injectable antihyperglycemic agents and/or insulin).
2. Had an admission for CF exacerbation less than 2 weeks prior to staring the medication. This will be defined as requiring new IV or PO antibiotics different than those used in maintenance therapy.
3. Is currently taking oral glucocorticoids or has been on oral or IV glucocorticoids in the past 2 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Glucose | 3 months
  This will be compared from baseline to 3 months after starting the medication
Change in Fasting Glucose | 6 months
  This will compare baseline to 6 months after starting the medication

SECONDARY OUTCOMES:
Genetic risk score | 6 months
  We will examine how the OGTT data is dependent on genotype at variants associated with type 2 diabetes using a genetic risk score
Pulmonary function test (PFT) FEV1 measurements | 6 months
  We will compare how PFT measurement of FEV1 are related to changes in OGTT
Change in Fasting Insulin | 3 months
  This will be compared from baseline to 3 months after starting the medication
Change in Fasting Insulin | 6 months
  This will be compared from baseline to 6 months after starting the medication

CONTACTS AND LOCATIONS:
Overall Officials: Jose Florez, MD, PhD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Wainwright CE, Elborn JS, Ramsey BW, Marigowda G, Huang X, Cipolli M, Colombo C, Davies JC, De Boeck K, Flume PA, Konstan MW, McColley SA, McCoy K, McKone EF, Munck A, Ratjen F, Rowe SM, Waltz D, Boyle MP; TRAFFIC Study Group; TRANSPORT Study Group. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Jul 16;373(3):220-31. doi: 10.1056/NEJMoa1409547. Epub 2015 May 17. PMID 25981758
- [Background] Bellin MD, Laguna T, Leschyshyn J, Regelmann W, Dunitz J, Billings J, Moran A. Insulin secretion improves in cystic fibrosis following ivacaftor correction of CFTR: a small pilot study. Pediatr Diabetes. 2013 Sep;14(6):417-21. doi: 10.1111/pedi.12026. Epub 2013 Mar 13. PMID 23952705